CLINICAL TRIAL: NCT06170177
Title: Bladder Archive: Observational Study on the Quality of Life and Pathological State in Patients Who Underwent Radical Cystectomy
Brief Title: Study on the Quality of Life and Pathological State in Patients Who Underwent Radical Cystectomy
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco Montorsi, Professor, IRCCS San Raffaele
Other Study IDs: 2012/Vescica
Record Dates: First submitted 2023-10-16; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Muscle Invasive Bladder Urothelial Carcinoma; Bladder Cancer TNM Staging; Bladder Cancer Stage IIa; Bladder Cancer Stage IIb; Bladder Cancer Stage IV; Bladder Leiomyosarcoma; Bladder Cancer; Bladder Cancer Stage II; Bladder Cancer Stage IIIa; Bladder Cancer Stage IIIb; Bladder Cancer Stage IIIc; Bladder Urothelial Carcinoma; Progression, Disease; Urinary Diversion; Neobladder; Radical Cystectomy
Keywords: Radical Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Disease Progression | interventions — Cystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent radical cystectomy
  Interventions: Procedure: Radical Cystectomy

INTERVENTIONS:
Procedure: Radical Cystectomy — A radical cystectomy is an operation to remove the whole bladder

SUMMARY:
Observational study on the quality of life and pathological state of patients underwent radical cystectomy.

DETAILED DESCRIPTION:
Each patient will be followed for approximately 10 years starting from the date of surgery. The patient may be contacted for yearly follow-up through one of the preferred methods indicated (phone call, email or home address) which will be carried out by the staff of the Urology Department. The data for each patient will then be transferred to the database itself. The data collected will be handled following the most strict GCPs and privacy norms.

The data entered will concern:

* period before hospitalization (symptoms, clinical data) and completion of a pre-surgery questionnaire
* hospitalization period with all its related data
* questionnaires relating to quality of life which will be administered to the patient once a year according to the preferred method expressed by the patient in the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* subjects underwent radical cystectomy
* > 18 years old
* Ability to read and sign the informed consent

Exclusion Criteria:

* Age <18 years
* Inability to read and sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with muscle-invasive bladder cancer underwent radycal cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2013-02-04 (Actual); Primary Completion 2063-02 (Estimated); Study Completion 2063-02 (Estimated)

PRIMARY OUTCOMES:
obtain health benefit for the patients themselves and for future patients underwent radical cystectomy | Baseline and Follow-up. 1 Annual follow-up until the patient decides to stop providing follow-up responses or until the date of death from any cause.
  All patients, before underwent radical cystectomy, receive a diary in which we ask a detailed clinical history of the patient with their symptoms, diagnosis and previous urological e non urological treatments performed before the operation. A detailed intraoperative, postoperative and follow-up clinical history.
improve the patient's scientific knowledge and develop new procedures for the diagnosis and treatment of the patient | Baseline and Follow-up. 1 Annual follow-up until the patient decides to stop providing follow-up responses or until the date of death from any cause.
  Through the collection of a detailed clinical history of the patient in which themselves report symptoms, diagnosis and previous urological and non-urological treatments and also through the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Montorsi, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No